CLINICAL TRIAL: NCT02405546
Title: Effect of 90° Degree Counterclockwise Rotation of the Endotracheal Tube on Its Advancement Through the Larynx During Nasal Fiberoptic Intubation in Children: A Randomized and Blinded Study
Brief Title: ETT Rotation During Nasal Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Dinesh Choudhry, MD, FRCA, Nemours Children's Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DC0001
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Dental Caries
Keywords: Nasal intubation; Counterclockwise rotation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-Rotated Technique (Group R) (Experimental): 90° counterclockwise rotation of bevel of ETT
  Interventions: Other: Pre-Rotated (Group R)
- No rotation (Active Comparator): No rotation of bevel of ETT
  Interventions: Other: No pre-rotation

INTERVENTIONS:
Other: Pre-Rotated (Group R) — In group R, placement of ETT over the FOS was done with 90° CCR from the beginning so that the bevel of the ETT faced posteriorly before it was advanced through the larynx.
  Other Names: 90° CCR
  Arms: Pre-Rotated Technique (Group R)
Other: No pre-rotation — ETT was not pre-rotated but rotated only if necessary
  Arms: No rotation

SUMMARY:
A nasal endotracheal tube (ETT) is routinely placed in children and a fiberoptic scope (FOS) is commonly used for this purpose. Resistance to the passage of ETT is frequently encountered as it is advanced over the FOS for placement into the trachea, since it gets hung up on structures of the laryngeal inlet. The aim of the investigators study performed on forty children divided in two groups was to study in the pediatric population, whether a 90° counterclockwise rotation (CCR) of the ETT prior to advancing through the larynx, by nasal approach, prevents it from getting hung up at the laryngeal inlet.

DETAILED DESCRIPTION:
A nasal endotracheal tube (ETT) is routinely placed in children and a fiberoptic scope (FOS) is commonly used for this purpose. Resistance to the passage of ETT is frequently encountered as it is advanced over the FOS for placement into the trachea, since it gets hung up on structures of the laryngeal inlet. The aim of the investigators study performed on forty children divided in two groups was to study in the pediatric population, whether a 90° counterclockwise rotation (CCR) of the ETT prior to advancing through the larynx, by nasal approach, prevents it from getting hung up at the laryngeal inlet.Following the approval of Nemours Institutional Review Board, and informed consent, forty healthy children were included in the study.

All children were randomly assigned to one of two groups using a computer generated numbers table. Group-S (Standard technique): It involved placement of ETT over the FOS with bevel of the ETT facing left as is routinely done Group-R (pre-Rotated technique): It involved placement of ETT over the FOS with 90° CCR from the beginning so that the bevel of the ETT faced posteriorly.

All children received midazolam premedication prior to coming to the operating room and were anesthetized by a standard technique using mask induction with oxygen, nitrous oxide and sevoflurane. Intravenous line was placed and rocuronium 0.4 mg/kg body weight was then administered to achieve muscle relaxation. Oxymetazoline hydrochloride lotion (Afrin) was sprayed in both nostrils to achieve nasal mucosal decongestion and the ETT of appropriate size for that age was used for nasotracheal intubation. Small FOS (Olympus LF-P; 2.2 mm diameter) was used for cuffed ETT (MallinckrodtTM; Covidien) sizes 4.5 mm ID and under and larger FOS (Olympus LF-DP; 3.1 mm diameter) was used for cuffed ETT (MallinckrodtTM; Covidien) sizes 5 mm ID and over. ETT was mounted on a FOS and secured near the proximal end close to the eyepiece. With head maintained in neutral position, a lubricated FOS was then advanced through the right or left nostril (the one that looked bigger) into the larynx and once in the trachea, the lubricated ETT was advanced over it.

An unblinded anesthesia attending associated with the study prepared the FOS and ETT according to the randomization, and advanced the FOS into the trachea and the ETT into the posterior pharynx. The anesthesia provider advancing the ETT was always one of the trainees: student nurse anesthetists (SRNA) or resident who was not a part of the study and was blinded to whether or not the ETT has been rotated 90°counterclockwise. The attending member of the research team observed as the ETT was advanced by the trainee and made a note of whether or not the ETT got hung up. If it did, the research team member withdrew the ETT 2 cm, rotated it 90° CCR, and allowed the trainee to advance the ETT one or more times, noting the results.

Following parameters would be measured:

Demographic data: age, weight, sex, nostril used and FOS size used; Whether or not ETT got hung-up at the laryngeal inlet, Whether or not 90° counterclockwise rotation was helpful with ETT advancement through the larynx and number of attempts needed to successfully advance the ETT after the 90° CCR.

Definition of resistance to tube advancement (hung-up ETT):

Steady but gentle force is generally needed to advance an ETT over the FOS, first through the nose and then into the trachea through the larynx. If the ETT were to pass smoothly no change in force is generally needed as it goes through the larynx. During advancement over the FOS, if ETT came to an abrupt stop and then the same steady force was insufficient to advance the ETT through the larynx it was defined as "hung up". If sudden resistance to passage through the larynx was encountered indicating that the ETT is hung up at the laryngeal inlet, it was then withdrawn about 2 cm, rotated 90° counterclockwise and readvanced through the larynx and observation was made if CCR maneuver leads to smoother passage of the ETT through the larynx into the trachea without it getting hung-up.

Statistical analysis: The data will be analyzed in the following manner: Nominal data such as gender, nostril used and FOS size compared between the groups using Fisher's exact test and numeric data such as age and weight with independent sample t-test. Outcome data such as presence or absence of resistance due to hung up ETT will be analyzed with Chi square while number of attempts will be analyzed with t-test. Significance was assumed at P< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 and 2
* Between 2 up to 18 years of age
* Normal airway anatomy
* scheduled for oral rehabilitation procedure

Exclusion Criteria:

* Children less than 2 years of age
* Abnormal airway and facial anatomy
* American Society of Anesthesiologists physical status 3 and 4
* Coagulation disorders were excluded from the study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Whether or not ETT got hung-up at the laryngeal inlet, the 90° CCR. | Outcome will be measured Immediately
  Definition of resistance to tube advancement (hung-up ETT): Steady but gentle force is generally needed to advance an ETT over the FOS, first through the nose and then into the trachea through the larynx. If the ETT were to pass smoothly no change in force is generally needed as it goes through the larynx. During advancement over the FOS, if ETT came to an abrupt stop and then the same steady force was insufficient to advance the ETT through the larynx it was defined as "hung up".

SECONDARY OUTCOMES:
Whether or not 90° counterclockwise rotation was helpful with ETT advancement through the larynx and number of attempts needed to successfully advance the ETT after | Outcome will be measured Immediately after the rotation is performed

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh K Choudhry, MD, FRCA, Principal Investigator — Nemours, DuPont Hospital for Children, Wilmington Deleware 19803
Locations (1):
- Nemours DuPont Hospital for Children, Wilmington, Delaware, United States

REFERENCES:
- [Background] Johnson DM, From AM, Smith RB, From RP, Maktabi MA. Endoscopic study of mechanisms of failure of endotracheal tube advancement into the trachea during awake fiberoptic orotracheal intubation. Anesthesiology. 2005 May;102(5):910-4. doi: 10.1097/00000542-200505000-00008. PMID 15851876
- [Background] Maktabi MA, Hoffman H, Funk G, From RP. Laryngeal trauma during awake fiberoptic intubation. Anesth Analg. 2002 Oct;95(4):1112-4, table of contents. doi: 10.1097/00000539-200210000-00061. PMID 12351306
- [Background] Ovassapian A, Yelich SJ, Dykes MH, Brunner EE. Fiberoptic nasotracheal intubation--incidence and causes of failure. Anesth Analg. 1983 Jul;62(7):692-5. No abstract available. PMID 6859572
- [Background] Brull SJ, Wiklund R, Ferris C, Connelly NR, Ehrenwerth J, Silverman DG. Facilitation of fiberoptic orotracheal intubation with a flexible tracheal tube. Anesth Analg. 1994 Apr;78(4):746-8. doi: 10.1213/00000539-199404000-00022. PMID 8135395
- [Background] Randell T, Hakala P, Kytta J, Kinnunen J. The relevance of clinical and radiological measurements in predicting difficulties in fibreoptic orotracheal intubation in adults. Anaesthesia. 1998 Dec;53(12):1144-7. doi: 10.1046/j.1365-2044.1998.00612.x. PMID 10193214
- [Background] Hakala P, Randell T. Comparison between two fibrescopes with different diameter insertion cords for fibreoptic intubation. Anaesthesia. 1995 Aug;50(8):735-7. doi: 10.1111/j.1365-2044.1995.tb06108.x. PMID 7645711
- [Background] Asai T, Shingu K. Difficulty in advancing a tracheal tube over a fibreoptic bronchoscope: incidence, causes and solutions. Br J Anaesth. 2004 Jun;92(6):870-81. doi: 10.1093/bja/aeh136. Epub 2004 Apr 30. No abstract available. PMID 15121723
- [Background] Kristensen MS, Moller J. Airway management behaviour, experience and knowledge among Danish anaesthesiologists--room for improvement. Acta Anaesthesiol Scand. 2001 Oct;45(9):1181-5. doi: 10.1034/j.1399-6576.2001.450921.x. PMID 11683672
- [Background] Schwartz D, Johnson C, Roberts J. A maneuver to facilitate flexible fiberoptic intubation. Anesthesiology. 1989 Sep;71(3):470-1. doi: 10.1097/00000542-198909000-00038. No abstract available. PMID 2774282
- [Background] Aoyama K, Takenaka I. Markedly displaced arytenoid cartilage during fiberoptic orotracheal intubation. Anesthesiology. 2006 Feb;104(2):378-9; author reply 379-80. doi: 10.1097/00000542-200602000-00032. No abstract available. PMID 16436865